CLINICAL TRIAL: NCT00362102
Title: A Multi-center, Open Label, Non-randomized, Phase II Study to Assess the Activity and Safety of Cetuximab Plus Irinotecan in Subjects With EGFR-detectable Metastatic Colorectal Carcinoma
Brief Title: A Phase II Study of Cetuximab Plus Irinotecan in Patients With EGFR-detectable Metastatic Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-259
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Carcinoma
Keywords: EGFR-detectable metastatic colorectal carcinoma with documented progressive disease to irinotecan-based chemotherapy and failure
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

INTERVENTIONS:
Drug: Cetuximab

SUMMARY:
To evaluate the response rate of cetuximab plus irinotecan combination therapy in subjects with EGFR-detectable metastatic colorectal carcinoma who have documented progressive disease to irinotecan-based chemotherapy and who have failed (progressive disease or intolerance) previous oxaliplatin-based and fluoropyrimidine-based chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have surgically unresectable metastatic colorectal carcinoma.
* The subjects who have received and failed Ilinotecan, oxaliplatin and fluoropyrimidine-based chemotherapy
* ECOG PS 0-2

Exclusion Criteria:

* Subjects with symptomatic cerebral metastasis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Response according to the RECIST criteria accessed every 6 weeks

SECONDARY OUTCOMES:
Time to progression, duration of achieved response, and the disease control rate will be accessed in all patients who received Cetuximab. The worst toxicity grades per patients will be tabulated for adverse events and laboratory measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company

REFERENCES:
- [Result] Tahara M, Shirao K, Boku N, Yamaguchi K, Komatsu Y, Inaba Y, Arai T, Mizunuma N, Satoh T, Takiuchi H, Nishina T, Sakata Y. Multicenter Phase II study of cetuximab plus irinotecan in metastatic colorectal carcinoma refractory to irinotecan, oxaliplatin and fluoropyrimidines. Jpn J Clin Oncol. 2008 Nov;38(11):762-9. doi: 10.1093/jjco/hyn102. Epub 2008 Oct 4. PMID 18836202